CLINICAL TRIAL: NCT04417829
Title: The Impact of Transcatheter Aortic Valve Implantation on Left Ventricular Structure, Function and Outcome in Patients With Aortic Stenosis
Brief Title: Transcatheter Aortic Valve Implantation in Western NORway
Acronym: TAVI-NOR
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/33814/REK vest
Record Dates: First submitted 2020-05-26; First posted 2020-06-05 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2020-05

CONDITIONS: Aortic Stenosis; Hypertension
Keywords: Aortic stenosis; Echocardiography; Transcutaneous aortic valve implantation; Left ventricular dysfunction; Left ventricular hypertrophy; Mortality
MeSH Terms: conditions — Aortic Valve Stenosis; Hypertension; Ventricular Dysfunction, Left; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Only one arm (intervention=TAVI): There is not control group/arm for comparison.
  Interventions: Device: Biological prosthesis in the aortic valve

INTERVENTIONS:
Device: Biological prosthesis in the aortic valve — Transcatheter aortic valve implantation of bioprosthesis in patients with severe symptomatic aortic stenosis (clinically indicated)

SUMMARY:
A prospective study of 600 patients with severe aortic stenosis (AS) and symptoms who underwent TAVI at the Haukeland university hospital, Bergen, Norway.

DETAILED DESCRIPTION:
A prospective study of 600 patients with severe aortic stenosis (AS) and symptoms who underwent TAVI at the Haukeland university hospital, Bergen, Norway between January 2012 and July 2019.

Demographics, clinical data including cardiovascular risk factors, arterial and echocardiographic parameters were prospectively collected. The data on all-cause mortality will be collected. Echocardiograms (immediate before TAVI, at discharge after TAVI and at 6-12 months follow-up) will be analyzed. The main scientific objectives are:

To assess survival benefits of TAVI according to baseline risk profile. To determine the echocardiographic predictors of left ventricular mass regression and left ventricular function recovery.

To evaluate global LV load (Zva=valvular-arterial impedance) following TAVI. To assess the impact of various types of blood pressure responses immediately after TAVI on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Hemodynamically severe aortic stenosis and symptoms
2. A decision of TAVI by Heart team
3. Patients undergoing TAVI (transcatheter aortic valve implantation)
4. Life expectancy > 1-2 years

Exclusion Criteria:

1. Sever frailty
2. Severly reduced cognitive function
3. Multiple comorbid conditions
4. Technically not suited for TAVI

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 600 patients with moderate or severe aortic stenosis of any etiology, and symptoms, where aortic valve intervention was clinially indicated. All patients underwent a successful TAVI (transcatheter aortic valve implantation).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
The impact of TAVI on all-cause mortality | From January 2012 to Mai 2020 (date for assesment vital status) + prolonged follow-up (up to 10 years)
  To assess the long-term survival benefits of TAVI
The impact of TAVI on left ventriclar mass and hypertrophy regression | From January 2012 to follow-up echo (6-12 months following TAVI)
  To assess whether removal of valve stenosis by TAVI leads to regression of left ventricular mass (grams).
The impact of TAVI on left ventricular function recovery | From January 2012 to to follow-up echo (6-12 months following TAVI)
  To assess improvement in systolic function (increase in ejection fraction) following TAVI
The impact of TAVI on arterial load (systemic arterial stiffness and arterial compliance). | From January 2012 to to follow-up echo (6-12 months following TAVI)
  To assess improvement in echocardiographic arterial stiffness and arterial compliance and global left ventricular load (Zva=valvular-arterial impedance) following TAVI.

CONTACTS AND LOCATIONS:
Overall Officials: Sahrai Saeed, MD.Ph.D., Principal Investigator — Department of Heart Disease Haukeland University Hospital, Begen, Norway

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers

REFERENCES:
- [Derived] Wasim D, Ali AM, Bleie O, Packer EJS, Eriksen E, Keilegavlen H, Rajani R, Rotevatn S, Saeed S. Prevalence and predictors of permanent pacemaker implantation in patients with aortic stenosis undergoing transcatheter aortic valve implantation: a prospective cohort study. BMJ Open. 2025 Feb 7;15(2):e093073. doi: 10.1136/bmjopen-2024-093073. PMID 39920059
- [Derived] Mohamed Ali A, Wasim D, Loland KH, Rotevatn S, Bleie O, Saeed S. Impact of transcatheter aortic valve implantation on left ventricular function recovery, mass regression and outcome in patients with aortic stenosis: protocol of the TAVI-NOR prospective study. BMJ Open. 2021 Jan 20;11(1):e039961. doi: 10.1136/bmjopen-2020-039961. PMID 33472776